CLINICAL TRIAL: NCT06314126
Title: Evaluation of D-Chiro-Inositol Treatment in Women With Endometriosis
Acronym: ENDO-DCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Principal Investigator, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDO-DCI
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Endometriosis
Keywords: D-Chiro-Inositol; Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and investigators will be masked to the treatment allocation. Treatment pills and placebo pills will be the same in shape, taste, color, and size.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-Chiro-Inositol (Experimental): Patients will receive oral D-Chiro-Inositol.
  Interventions: Dietary Supplement: D-Chiro-Inositol
- Placebo (Placebo Comparator): Patients will receive oral placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: D-Chiro-Inositol — Patients in the experimental group will receive 1200 mg of oral D-Chiro-Inositol per day.
  Arms: D-Chiro-Inositol
Other: Placebo — Patients in the control group will receive 1200 mg of placebo per day.
  Arms: Placebo

SUMMARY:
To date, the treatment for endometriosis is represented by the surgical removal of the lesions. Nonetheless, in the years following surgery, the lesions can recur, often due to excessive estrogen production. To balance estrogen, progestin- or estrogen-progestin-based medications are generally prescribed. On the other hand, progestins and estrogen-progestins act as contraceptives, preventing the onset of a pregnancy. At the same time, these can have side effects that can affect up to 30% of patients. For these and other reasons, some women refuse therapy with progestins or estrogen-progestins, preferring to resort to no treatment.

Considering the need to research effective molecules in the prevention of relapses that can maintain fertility and avoid unwanted effects, the research focuses on natural molecules, well tolerated by the body.

D-Chiro-Inositol (DCI) is a polyol normally present in human cell membranes, where, from a metabolic point of view, it acts as a second messenger of insulin, while from a hormonal point of view, it exerts an on the biosynthesis of androgens. This effect on steroidogenesis can be attributed to more than one mechanism. In the ovary, DCI stimulates direct testosterone production. Furthermore, it stimulates the accumulation of testosterone by reducing the activity of the aromatase enzyme, responsible for the conversion of androgens into estrogens. Considering the responsiveness of endometriosis to estrogens, and that these constitute a risk factor for recurrences following surgical removal, the use of DCI could be interesting from a clinical point of view.

The study plans to verify whether D-Chiro-Inositol dietary supplementation can be effective in reducing systemic estrogen levels in women with endometriosis, thus also reducing the risk of relapses and associated symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Women affected by endometriosis (regardless of the stage)

Exclusion Criteria:

* Treatment with hormones in the previous three months or during the study
* Treatment with Inositol and/or other insulin-sensitizers in the previous three months
* Obesity
* Diabetes
* Cancer (any site/stage)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Estradiol | At the 3° day of the menstrual cycle before to start the study, after one month, after three months, after six months from the enrollment
  Serum estradiol level by peripheral blood test

SECONDARY OUTCOMES:
Pelvic pain | At the 3° day of the menstrual cycle before to start the study, after one month, after three months, after six months from the enrollment
  Pelvic pain measured as visual analog scale (VAS), from 0 (no pain) to 10 (maximal perceived pain).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — University of Palermo; Pietro Serra, M.D., Study Chair — University of Palermo; Giuseppe Mascellino, M.D., Study Chair — University of Palermo; Andrea Etrusco, M.D., Study Chair — University of Palermo
Locations (1):
- "Paolo Giaccone" Hospital, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No